CLINICAL TRIAL: NCT02376998
Title: Endovascular Repair for Acute Traumatic Transection of the Descending Thoracic Aorta
Brief Title: Endovascular Repair for the Descending Thoracic Aorta
Acronym: ERRATA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Prof. Raffaele Serra, MD, Ph.D., Prof. Raffaele Serra, University of Catanzaro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERRATASTUDY
Record Dates: First submitted 2015-02-12; First posted 2015-03-03 (Estimated); Results first posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-08

CONDITIONS: Aorta Thoracic; Traumatic Rupture
Keywords: Thoracic Aorta; Trauma; Endovascular
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Valiant™ endoluminal procedure (Experimental): Data from early and long term complications following endoluminal stent-graft placement for thoracic endovascular aortic repair (TEVAR) procedure (Valiant™ endoluminal procedure) will be collected.
  Interventions: Device: Valiant™ endoluminal procedure

INTERVENTIONS:
Device: Valiant™ endoluminal procedure — Thoracic endovascular aortic repair with Endoluminal stent-graft placement (Valiant™ endoluminal stent-graft systems (Medtronic Inc., Santa Rosa, CA, USA) will be performed as follows:
  The diameter of the stent graft will be calculated from the largest diameter of the proximal/distal neck with an oversizing factor of 10-20%. The procedures will be done with local or general anaesthesia in case of unstable pre-operative hemodynamic conditions.
  After the procedure will be completed, a digital subtraction angiography and echocardiography with color-flow mapping were performed to verify the correct positioning of the stent and to detect any primary endoleak.

SUMMARY:
Most blunt aortic injuries occur in the proximal proximal descending aorta causing acute transection of this vessel. Generally, surgical repair of the ruptured segment of aorta is associated with high rates of morbidity and mortality and in this view endovascular treatment seems to be a valid and safer alternative. Aim of this study is to review the experience of a single center with endovascular approach for the treatment of acute traumatic rupture of descending thoracic aorta

DETAILED DESCRIPTION:
From April 2002 to November 2014, patients referred to our Department with a diagnosis of acute transection of thoracic aorta will be studied by preoperative Computed Tomography (CT) evaluation in order to perform thoracic endovascular aortic repair (TEVAR) with left subclavian artery coverage. Then patients will be followed up with clinical and instrumental (CT, Duplex ultrasound) controls at discharge, 1, 3 and 6 months and yearly thereafter. We will evaluate the presence of major and minor neurological complications, episodes of left arm claudication, cardiovascular, respiratory and bleeding complications. Furthermore we will evaluate the technical success of the technique evaluating the onset of failure, collapse, leak or distal migration of the graft.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of acute transection of thoracic aorta;
* a time frame range from trauma of 1-10 hours.

Exclusion Criteria:

* Patients who do not fall into the above categories

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2002-11; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serra R, de Franciscis S, Grande R, Butrico L, Perri P, Indolfi C, Mastroroberto P. Endovascular repair for acute traumatic transection of the descending thoracic aorta: experience of a single centre with a 12-years follow up. J Cardiothorac Surg. 2015 Nov 21;10:171. doi: 10.1186/s13019-015-0388-5. PMID 26590963

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Acute Transection of Thoracic Aorta: Patients with a diagnosis of acute transection of thoracic aorta.
Period: Overall Study
Arm/Group | Patients With Acute Transection of Thoracic Aorta
Started | 20
Completed | 11
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Acute Transection of Thoracic Aorta
Number analyzed (Participants) | 11
Age, Continuous [Mean (Full Range); unit: years] | 36.9 [18 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Region of Enrollment [Number; unit: participants]
  Italy | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Adverse Events
Description: Evaluation of mortality, renal failure, cerebrovascular accident.
Time Frame: from hospital discharge to 1 month after the procedure
Population: No serious adverse events recorded
Measure: Number; unit: number of serious adverse events
Groups:
- Patients With Acute Transection of Thoracic Aorta: Patients with a diagnosis of acute transection of thoracic aorta. Mortality 0%
Arm/Group | Patients With Acute Transection of Thoracic Aorta
Number analyzed (Participants) | 11
number of serious adverse events | 0

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Valiant™ Endoluminal Procedure: Data from early and long term complications following endoluminal stent-graft placement for thoracic endovascular aortic repair (TEVAR) procedure (Valiant™ endoluminal procedure) will be collected.
  Valiant™ endoluminal procedure: Thoracic endovascular aortic repair with Endoluminal stent-graft placement (Valiant™ endoluminal stent-graft systems (Medtronic Inc., Santa Rosa, CA, USA) will be performed as follows:
  The diameter of the stent graft will be calculated from the largest diameter of the proximal/distal neck with an oversizing factor of 10-20%. The procedures will be done with local or general anaesthesia in case of unstable pre-operative hemodynamic conditions.
  After the procedure will be completed, a digital subtraction angiography and echocardiography with color-flow mapping were performed to verify the correct positioning of the stent and to detect any primary endoleak.
Arm/Group | Valiant™ Endoluminal Procedure
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No